CLINICAL TRIAL: NCT01517074
Title: A Phase I/II Study to Investigate Subconjunctival Sirolimus for the Treatment of Active Autoimmune Non-Necrotizing Anterior Scleritis
Brief Title: Sirolimus Injections for Autoimmune Scleritis
Acronym: ISAS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120057; 12-EI-0057
Record Dates: First submitted 2012-01-24; First posted 2012-01-25 (Estimated); Results first posted 2014-06-10 (Estimated); Last update posted 2020-06-19 (Actual); Status verified 2016-08

CONDITIONS: Scleritis
Keywords: Sirolimus; Scleritis; Autoimmune Scleritis
MeSH Terms: conditions — Scleritis | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sirolimus (Experimental): Participants will receive a15 μL (660 μg) subconjunctival injection of sirolimus in the study eye at baseline if a single quadrant or two adjacent quadrants are involved. If greater than two quadrants are involved (i.e., 3 or 4 quadrant involvement) or two non-adjacent quadrants are involved, two 15 μL (660 μg) injections will be given in two quadrants 180 degrees apart (total dose of 30 μL or 1,320 μg). Participants that still demonstrate active inflammation (incomplete or no response to initial injection) or experience a flare-up (as defined by a ≥1-step increase in scleral inflammation) after the initial injection will be eligible for a re-injection in the study eye at or after Week 4 (not to exceed a dose of 1,320 μg per eye within an eight-week period).
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Subconjunctival injection
  Other Names: Rapamune®; rapamycin

SUMMARY:
Background:

Autoimmune scleritis is an inflammatory disease that affects the white outer part of the eye. It is associated with immune system disorders like rheumatoid arthritis. It can cause blindness in severe cases. Most treatments for scleritis involve steroid or immune-suppressing drugs, but these can cause side effects in the whole body.

Sirolimus is a drug used to help prevent transplant rejection. It helps prevent the immune system from attacking the body. Researchers want to try giving sirolimus injections into the eye to treat severe scleritis.

Objectives:

To see if sirolimus is a safe and effective treatment for autoimmune scleritis.

Eligibility:

Individuals at least 18 years of age with autoimmune scleritis in at least one eye that has not responded to standard treatments.

Design:

* Participants will be screened with a medical history, physical exam, and eye exam. Blood and urine samples will also be collected.
* One eye will be selected as the study eye to receive injections.
* Participants will have six study visits over 4 months (initial visit and weeks 2, 4, 8, 12, and 16). The injection will be given at the first visit. If the study eye responds to the treatment, participants may have injections in the other eye at the second visit.
* If there is still inflammation after the first injection, or if the scleritis improves but then returns, participants may have a second injection at Week 4.
* Injections will be monitored with blood tests and eye exams.
* Participants may have study visits and injections for up to 1 year if the injections seem to be working.

DETAILED DESCRIPTION:
OBJECTIVE:

Scleritis is a chronic, painful and potentially blinding inflammatory disease characterized by edema of the episcleral and scleral tissues and is commonly associated with systemic autoimmune disorders. Sirolimus suppresses cytokine-driven T-cell proliferation and thus, inhibits the production, signaling and activity of many growth factors relevant to scleritis. Subconjunctival sirolimus administration could reduce or eliminate the need for topical and/or systemic immunosuppressive drugs often taken with immunosuppressive disorders that could result in reduced morbidity. The study objective is to investigate the safety, tolerability and potential efficacy of subconjunctival sirolimus as a possible treatment for active, autoimmune, non-necrotizing, anterior scleritis.

STUDY POPULATION:

Five participants with active, autoimmune, non-necrotizing, anterior scleritis with scleral inflammatory grade ≥ 1+ in at least one quadrant will be initially enrolled. Participants must have a history of past flares requiring oral non-steroidal anti-inflammatory drugs (NSAIDS), or oral or topical corticosteroids or immunosuppressive medication. Up to seven participants may be enrolled, as up to two participants may be accrued to account for participants who withdraw from the study prior to receiving any investigational product.

DESIGN:

This is a phase I/II, single-center, open-label, non-randomized, prospective and uncontrolled pilot study to evaluate the safety and possible efficacy of subconjunctival sirolimus injections for active, autoimmune, non-necrotizing, anterior scleritis. If two eyes are active, the eye with worse inflammation will be injected first (study eye) at baseline followed two weeks later with injection of the second eye (fellow eye). If both eyes have equal inflammation, the study eye will be chosen at the physician's discretion after consultation with the participant. Participants that still demonstrate active inflammation or experience a flare-up after the initial study eye injection may be eligible for a re-injection at or after Week 4 (not to exceed a dose of 1,320 μg per eye within an eight-week period).

OUTCOME MEASURES:

The primary outcome is the number of participants who experience at least a 2-step reduction or reduction to grade 0 of scleral inflammation in the study eye according to a standardized photographic scleritis grading system developed at the National Eye Institute (NEI) by the Week 8 visit. Secondary outcomes include changes in visual acuity, step changes in scleral inflammation, the number of participants who experience a disease flare, the number of participants tapered from the standard immunosuppressive regimen after 16 weeks and, of the participants who experience a disease flare, the number of days to disease flare from baseline as well as the number of participants who require re-injection due to a flare. Safety outcomes include the number and severity of systemic and ocular toxicities and adverse events (AEs), the proportion of participants who experience vision loss ≥ 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters and the number of participants who experience a substantial rise in elevated intraocular pressure (IOP).

ELIGIBILITY:
INCLUSION CRITERIA:

1. Participant has the ability to understand and sign the informed consent document.
2. Participant is 18 years of age or older.
3. Participant has a diagnosis of active, autoimmune, non-necrotizing, anterior scleritis.
4. Participant, if currently taking immunosuppressive medications, is on a stable regimen of immunosuppressive medications (no increase and/or start of new immunosuppressive medications) over the last four weeks.
5. Participant has tried therapy such as oral non-steroidal anti-inflammatory drugs (NSAIDs), or oral or topical corticosteroids or immunosuppressive medication at any time in the past to control scleritis flares, or has intolerance or contraindications to these medications.
6. Participant is willing and able to comply with the study procedures.
7. Female participants of childbearing potential must not be pregnant or breast-feeding, have a negative pregnancy test at screening and must be willing to undergo pregnancy tests throughout the study.
8. Both female participants of childbearing potential and male participants able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse or must agree to practice two acceptable methods of contraception throughout the course of the study and for four months after the last investigational product injection. Acceptable methods of contraception include: hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring), intrauterine device, barrier methods (diaphragm, condom) with spermicide, or surgical sterilization (tubal ligation).

EXCLUSION CRITERIA:

1. Participant has a significant active intraocular infection in either eye that requires antibiotic treatment.
2. Participant has an active serious infection or a history of recurring serious infections such as human immunodeficiency virus (HIV) or syphilis that in the best medical judgment of the investigators would pose unnecessary risk to the participant.
3. Participant has active joint or systemic inflammation requiring immediate addition or increase in systemic anti-inflammatory medications.
4. Participant is taking systemic azole anti-fungal medication (e.g., ketoconazole, voriconazole, itraconazole).

STUDY EYE ELIGIBILITY CRITERIA:

The participant must have at least one eye meeting all inclusion criteria and none of the exclusion criteria listed below.

STUDY EYE INCLUSION CRITERIA:

1. Participant has anterior scleritis with greater than or equal to 1 plus in at least one quadrant of the study eye.
2. Participant has visual acuity in the study eye of 20/640 or better.
3. Participant agrees not to undergo elective intraocular surgery in the study eye (e.g., cataract extraction) for three months after the last injection.
4. Participant has not received a periocular or intravitreal injection in the study eye in the last six weeks.

STUDY EYE EXCLUSION CRITERIA:

1. Participant has necrotizing scleritis in the study eye.
2. Participant had intraocular surgery in the study eye in the last four weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hatice N Sen, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rothova A, Suttorp-van Schulten MS, Frits Treffers W, Kijlstra A. Causes and frequency of blindness in patients with intraocular inflammatory disease. Br J Ophthalmol. 1996 Apr;80(4):332-6. doi: 10.1136/bjo.80.4.332. PMID 8703885
- [Background] Jabs DA, Mudun A, Dunn JP, Marsh MJ. Episcleritis and scleritis: clinical features and treatment results. Am J Ophthalmol. 2000 Oct;130(4):469-76. doi: 10.1016/s0002-9394(00)00710-8. PMID 11024419
- [Background] Sen HN, Suhler EB, Al-Khatib SQ, Djalilian AR, Nussenblatt RB, Buggage RR. Mycophenolate mofetil for the treatment of scleritis. Ophthalmology. 2003 Sep;110(9):1750-5. doi: 10.1016/S0161-6420(03)00570-0. PMID 13129873
- [Result] Bhatt N, Dalal M, Tucker W, Obiyor D, Nussenblatt R, Sen HN. Subconjunctival sirolimus in the treatment of autoimmune non-necrotizing anterior scleritis: results of a phase I/II clinical trial. Am J Ophthalmol. 2015 Mar;159(3):601-6. doi: 10.1016/j.ajo.2014.12.009. Epub 2014 Dec 17. PMID 25526946
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-EI-0057.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sirolimus
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (15.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least 2-step Reduction or Reduction to Grade 0 of Scleral Inflammation in the Study Eye According to the National Eye Institute (NEI) Photographic Scleritis Grading System Within 8 Weeks Post-injection.
Description: The primary efficacy outcome was a 2-step reduction in scleritis grading out of a scale of 0 to 4+ (where 0.5+ is recognized as an ordinal step between 1+ and 0+).
  Scleral inflammation was graded following 10% Phenylephrine application with an ordinal scale of 0 (no scleral inflammation with complete blanching of vessels), 0.5+ (minimal/trace inflammation with localized pink appearance of the sclera around minimally dilated deep episcleral vessels), 1+ (mild inflammation with diffuse pink appearance of the sclera around mildly dilated deep episcleral vessels), 2+ (moderate inflammation with purplish pink appearance of the sclera with tortuous and engorged deep episcleral vessels), 3+ (severe inflammation with diffuse significant redness of sclera, the details of superficial and deep episcleral vessels can't be observed), and 4+ (necrotizing inflammation with diffuse redness of the sclera with scleral thinning and uveal show).
Time Frame: Baseline and Week 8
Measure: Number; unit: participants
Groups:
- Sirolimus: Participants will receive a 15 μL (660 μg) subconjunctival injection of sirolimus in the study eye at baseline if a single quadrant or two adjacent quadrants are involved. If > two quadrants are involved (i.e., 3 or 4 quadrant involvement) or two non-adjacent quadrants are involved, two 15 μL (660 μg) injections will be given in two quadrants 180 degrees apart (total dose of 30 μL or 1,320 μg).
  Participants that still demonstrate active inflammation (incomplete or no response to initial injection) or experience a flare-up (as defined by a ≥1-step increase in scleral inflammation) after the initial injection will be eligible for a re-injection in the study eye at or after Week 4 (not to exceed a dose of 1,320 μg per eye within an eight-week period).
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
participants | 5

2. Secondary Outcome: Number of Participants Who Experience a Disease Flare as Defined by a ≥ 1-step Increase in Scleral Inflammation
Description: Scleral inflammation was graded following 10% Phenylephrine application with an ordinal scale of 0 (no scleral inflammation with complete blanching of vessels), 0.5+ (minimal/trace inflammation with localized pink appearance of the sclera around minimally dilated deep episcleral vessels), 1+ (mild inflammation with diffuse pink appearance of the sclera around mildly dilated deep episcleral vessels), 2+ (moderate inflammation with purplish pink appearance of the sclera with tortuous and engorged deep episcleral vessels), 3+ (severe inflammation with diffuse significant redness of sclera, the details of superficial and deep episcleral vessels can't be observed), and 4+ (necrotizing inflammation with diffuse redness of the sclera with scleral thinning and uveal show)
Time Frame: Baseline and Week 52
Measure: Number; unit: participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
participants | 3

3. Secondary Outcome: Mean Change in Visual Acuity Via the Early Treatment Diabetic Retinopathy Study (ETDRS)
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
Time Frame: Baseline and Week 52
Population: Mean change in visual acuity at Week 52 from Baseline is presented for the study and fellow eyes for participants who completed follow-up through Week 52.
Measure: Mean (Standard Deviation); unit: letters read
Groups:
- Study Eye; Fellow Eye: Participants will receive a 15 μL (660 μg) subconjunctival injection of sirolimus in the study eye at baseline if a single quadrant or two adjacent quadrants are involved. If > two quadrants are involved (i.e., 3 or 4 quadrant involvement) or two non-adjacent quadrants are involved, two 15 μL (660 μg) injections will be given in two quadrants 180 degrees apart (total dose of 30 μL or 1,320 μg).
  Participants that still demonstrate active inflammation (incomplete or no response to initial injection) or experience a flare-up (as defined by a ≥1-step increase in scleral inflammation) after the initial injection will be eligible for a re-injection in the study eye at or after Week 4 (not to exceed a dose of 1,320 μg per eye within an eight-week period).
Arm/Group | Study Eye | Fellow Eye
Number analyzed (Participants) | 4 | 4
letters read | -0.25 (3.69) | -2.25 (2.06)

4. Secondary Outcome: Median Change in Visual Acuity Via the Early Treatment Diabetic Retinopathy Study (ETDRS)
Description: as for outcome 3
Time Frame: Baseline and Week 52
Population: Median change in visual acuity at Week 52 from Baseline is presented for the study and fellow eyes for participants who completed follow-up through Week 52.
Measure: Median (Full Range); unit: letters read
Arm/Group | Study Eye | Fellow Eye
Number analyzed (Participants) | 4 | 4
letters read | 0.00 [-5.00 to 4.00] | -2.50 [-4.00 to 0.00]

5. Secondary Outcome: Number of Participants Needing a Second Injection
Description: Participants that still demonstrate active inflammation (incomplete or no response to initial injection) or experience a flare-up (as defined by a ≥1-step increase in scleral inflammation) after the initial injection will be eligible for a re-injection in the study eye at or after Week 4 (not to exceed a dose of 1,320 μg per eye within an eight-week period).
Time Frame: Baseline and Week 52
Measure: Number; unit: participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
participants | 3

6. Secondary Outcome: Mean Number of Days Between the First Injection to the Second Injection
Description: For participants who demonstrate active inflammation (incomplete or no response to initial injection) or experience a flare-up (as defined by a ≥1-step increase in scleral inflammation) after the initial injection
Time Frame: Baseline and Week 52
Measure: Mean (Full Range); unit: Days
Arm/Group | Sirolimus
Number analyzed (Participants) | 3
Days | 65.3 [28 to 84]

7. Secondary Outcome: Number of Participants Who Experienced Ocular Toxicities
Time Frame: Baseline and Week 52
Measure: Number; unit: participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
participants | 2

8. Secondary Outcome: Number of Participants Who Experienced Systemic Toxicities
Time Frame: Baseline and Week 52
Measure: Number; unit: participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
participants | 0

9. Secondary Outcome: Number of Participants Who Tapered Off One or More Systemic Immunosuppressive Medications or Tapered Off Prednisone (≤10 mg) After Week 16
Description: Four (4) out of 5 participants were on immunosuppressive medications at enrollment.
Time Frame: Week 16 and Week 52
Measure: Number; unit: participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 4
participants | 1

10. Secondary Outcome: Proportion of Participants With Loss of ≥ 15 Early Treatment Diabetic Retinopathy Study (ETDRS) Letters
Description: as for outcome 3
Time Frame: Baseline to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Study Eye | Fellow Eye
Number analyzed (Participants) | 5 | 5
Participants | 0 | 1

11. Secondary Outcome: Number of Participants Who Experience a Substantial Rise in Elevated Intraocular Pressure (IOP)
Description: A substantial rise in intraocular pressure can be defined as ≥10 mmHg change in pressure.
Time Frame: Baseline and Week 52
Measure: Number; unit: participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
participants | 0

12. Secondary Outcome: Step Changes in Scleral Inflammation According to the Standardized Photographic Grading System Developed at National Eye Institute (NEI)
Description: as for outcome 2
Time Frame: Baseline and Week 52
Population: Scleral inflammation scores are presented at Baseline and Week 52 and the step change in scores at Week 52 from Baseline for participants who completed follow-up through Week 52.
Measure: Number; unit: score on a scale
Groups:
- Scleral Inflammation Score at Baseline; Scleral Inflammation Score at Week 52; Step Changes in Scleral Inflammation at Week 52 From Baseline: Participants will receive a 15 μL (660 μg) subconjunctival injection of sirolimus in the study eye at baseline if a single quadrant or two adjacent quadrants are involved. If > two quadrants are involved (i.e., 3 or 4 quadrant involvement) or two non-adjacent quadrants are involved, two 15 μL (660 μg) injections will be given in two quadrants 180 degrees apart (total dose of 30 μL or 1,320 μg).
  Participants that still demonstrate active inflammation (incomplete or no response to initial injection) or experience a flare-up (as defined by a ≥1-step increase in scleral inflammation) after the initial injection will be eligible for a re-injection in the study eye at or after Week 4 (not to exceed a dose of 1,320 μg per eye within an eight-week period).
Arm/Group | Scleral Inflammation Score at Baseline | Scleral Inflammation Score at Week 52 | Step Changes in Scleral Inflammation at Week 52 From Baseline
Number analyzed (Participants) | 4 | 4 | 4
score on a scale
  Participant 001: number analyzed (Participants) | 1 | 1 | 1
  Participant 001 | 3 | 0 | -4
  Participant 002: number analyzed (Participants) | 1 | 1 | 1
  Participant 002 | 1 | 0 | -2
  Participant 003: number analyzed (Participants) | 1 | 1 | 1
  Participant 003 | 3 | 0 | -4
  Participant 005: number analyzed (Participants) | 1 | 1 | 1
  Participant 005 | 3 | 0 | -4

ADVERSE EVENTS:
Time Frame: 52 Weeks
Arm/Group | Sirolimus
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=5)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=5)
Pneumonia (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Wisdom teeth removal (Surgical and medical procedures) | 1 (1)
Eye inflammation (Eye disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No